CLINICAL TRIAL: NCT00574769
Title: Phase Ib/II Evaluation of RAD001 With Docetaxel and Bevacizumab in Patients With Metastatic Androgen Independent Prostate Cancer
Brief Title: Safety Study & Effectiveness of Docetaxel With RAD001 and Bevacizumab in Men With Advanced Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-09-4; AVF3955s; CRAD001CUS2468
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: RAD001; mTOR inhibition; docetaxel; bevacizumab; adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer; prostate cancer; Metastatic, androgen independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Everolimus; Docetaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RAD001, Docetaxel, Bevacizumab

INTERVENTIONS:
Drug: RAD001, Docetaxel, Bevacizumab — RAD001 oral, 2.5 mg daily RAD001 oral, 5mg daily
  Bevacizumab infusion (IV), 15 mg/kg every 21 days
  Docetaxel infusion (IV), 75 mg/m^2 every 21 days
  Other Names: everolimus; Avastin; Taxotere

SUMMARY:
Prostate cancer is a common and important health issue. Although effective treatment is often available for localized disease, metastatic prostate cancer remains incurable. The initial treatment for metastatic prostate cancer often includes medical or surgical treatments that deprive the tumor of male hormones (androgens) required for growth. Although this treatment is successful for many patients, the cancer may eventually return in others. Recurrent prostate cancer may be treated with additional hormonal agents, but these agents usually do not result in long-term control of the disease. Eventually most patients with recurrent prostate cancer progress to a state where the cancer grows despite very low level of circulating male hormones known as androgen independent prostate cancer (AIPC).

DETAILED DESCRIPTION:
Patients will undergo a screening procedure to determine eligibility of trial. During the treatment period, the patient will be given docetaxel/bevacizumab on day 1 followed by RAD001 continuously on days 2-21 and this is called a treatment cycle. Patients will be able to continue to receive multiple treatment courses as long as the cancer does not get worse and the person does not develop other problems that would prevent him from staying in the study. The final part of the research is the study completion period which includes an end of treatment visit and subsequent follow-up visits. These visits take place whenever the research medication is stopped, even if it is stopped early. For the patient's safety, he/she should at least complete the end of treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Signed informed consent
* ECOG performance status: 0-2
* Histologically documented adenocarcinoma of the prostate
* Progressive disease despite androgen deprivation therapy. Progressive disease is defined as any one of the following:
* Measurable Disease: Objective evidence of increase > 20% in the sum of the longest diameters of target lesions from the time of maximal regression or the appearance of one or more new lesions (Modified RECIST Criteria)
* Bone Scan Progression: Appearance of one or more new lesions on bone scan attributable to prostate cancer
* PSA Progression: An elevated PSA (≥ 5 ng/ml) which has risen serially from baseline on two occasions each at least one week apart
* At least 4 weeks since any other hormonal therapy. Flutamide and megestrol acetate (any dose) must be discontinued at least 4 weeks prior to initiating treatment. Bicalutamide or nilutamide must be discontinued at least 6 weeks prior to initiating treatment. If improvement following antiandrogen withdrawal is noted, progression must be established using the criteria above. Androgen suppression should be continued
* ≥ 4 weeks since major surgery and fully recovered
* ≥ 8 weeks since high risk surgery and fully recovered
* ≥ 4 weeks since any prior radiation and fully recovered
* ≥ 6 weeks since the last dose of bone targeted radiopharmaceutical
* Men of child-bearing potential are required to use an effective means of contraception
* Required Initial Laboratory Values:

  * ANC ≥ 1500/µL
  * Platelet count ≥ 100,000/µL
  * Creatinine ≤ 1.5 x ULN
  * Bilirubin ≤ 1.5 x ULN
  * AST ≤ 1.5 x ULN
  * Urine protein to creatinine ratio < 1.0
  * Serum Testosterone ≤ 50 ng/dL (For patients who have not had bilateral orchiectomy.)

Exclusion Criteria:

* Prior treatment with cytotoxic chemotherapy for metastatic disease
* Prior treatment with anti-angiogenic agents, including thalidomide and bevacizumab
* Prior treatment with any investigational drug within 4 weeks of initiating treatment
* Prior treatment with an mTor inhibitor
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Known history of HIV seropositivity
* Known brain metastases (brain imaging is not required)
* Congestive heart failure
* Uncontrolled hypertension. Patients with history of hypertension must be well controlled (< 150/100) on a regimen of anti-hypertensive therapy
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Active bleeding diathesis or on oral anti-vitamin K medications (except low dose coumarin)
* Arterial thrombotic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), at any time
* History of unstable angina or angina requiring surgical or medical intervention in the past 12 months, or myocardial infarction (MI)
* Patients with clinically significant peripheral artery disease or any other arterial thrombotic event
* Significant vascular disease
* Other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study
* Proteinuria at screening as demonstrated by either
* Urine protein:creatinine (UPC) ratio ≥ 1.0 OR
* Urine dipstick for proteinuria ≥ 2+
* Serious or non-healing wound, ulcer or bone fracture
* Peripheral neuropathy ≥ grade 2
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Herbal medications and food supplements must be discontinued before registration. Patients may continue on daily vitamins and calcium supplements
* History of noncompliance to medical regimens
* Unwilling to or unable to comply with the protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-02-17 (Actual); Primary Completion 2016-02-17 (Actual); Study Completion 2017-02-17 (Actual)

PRIMARY OUTCOMES:
Establish a maximal tolerated or optimal biologic dose of RAD001 in combination with docetaxel/bevacizumab | After the last patient in the cohort has completed at least two cycles of RAD001/docetaxel/bevacizumab

SECONDARY OUTCOMES:
Evaluate the efficacy of RAD001 in combination with docetaxel/bevacizumab as determined by best overall response and progression-free survival in patients with advanced prostate cancer. | overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell E Gross, MD, Ph.D, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Westside Prostate Cancer Center, University of Southern California, Beverly Hills, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California